CLINICAL TRIAL: NCT04791878
Title: A Phase I Study of Adult Allogeneic Bone Marrow Derived Mesenchymal Stem Cells for Pediatric Perianal Fistulizing Crohn's Disease
Brief Title: Study of Mesenchymal Stem Cells for Pediatric Perianal Fistulizing Crohn's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amy Lightner (Other)
Responsible Party: Sponsor-Investigator, Amy Lightner, MD, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-134
Record Dates: First submitted 2021-03-06; First posted 2021-03-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Perianal Fistula Due to Crohn's Disease (Disorder)
Keywords: perianal; fistula; pediatric; crohn's disease
MeSH Terms: conditions — Fistula; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mesenchymal stem cells (Experimental): allogeneic bone marrow derived mesenchymal stem cells
  Interventions: Drug: Mesenchymal stem cells

INTERVENTIONS:
Drug: Mesenchymal stem cells — Direct injection of 75 million allogeneic bone marrow derived mesenchymal stem cells at baseline and again after 3 months if not completely healed

SUMMARY:
This study plans to enroll 10 patients aged 13-17 years of age with refractory perianal fistulizing disease. Patients will be treated by direct injection to the fistula tract(s) with 75 million allogeneic bone marrow derived mesenchymal stem cells at baseline and again after 3 months if not completely healed.

DETAILED DESCRIPTION:
Crohn's disease (CD), a chronic transmural inflammatory disease of the gastrointestinal tract, continues to increase in incidence for unknown reasons. According to population based studies, at least 26% of patients with CD will develop perianal fistulas in the first two decades following diagnosis, particularly those with colonic and rectal involvement. These patients experience significant morbidity due to pain, persistent drainage, recurrent perianal sepsis, and ongoing need to access medical care resulting in increased costs and impaired quality of life. Onset of Crohn's disease in childhood is associated with even more aggressive perianal fistula development, with fistulas occurring in as many as 20-31% of children within 5-7 years after Crohn's disease diagnosis. Based on national estimates of pediatric Crohn's disease prevalence, this suggests that there are more than 10,000 children with perianal fistulas due to Crohn's disease in the United States.

This study plans to enroll 10 patients (aged 13-17 years) with refractory perianal fistulizing disease. The next step in management for these patients would be a mucosal tissue flap, temporary stoma, or proctectomy with permanent ostomy.

Patients will be treated by direct injection of 75 million allogeneic bone marrow derived mesenchymal stem cells at baseline and again after 3 months if not completely healed. Patients will be followed for a total of 12 months post initial injection.

ELIGIBILITY:
Inclusion Criteria

1. Males and females aged 13-17 with a diagnosis of Crohn's disease for at least six months duration.
2. Single and Multi-tract Perianal fistula, with or without previous failed surgical repair.
3. Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
4. Ability to comply with protocol
5. Competent and able to provide written informed consent
6. Concurrent Crohn's-related therapies with stable doses corticosteroids, 5- ASA drugs, immunomodulators, anti-TNF therapy, anti-integrin and anti-interleukin therapies are permitted.
7. Agree to use birth control or abstinence to avoid pregnancy during the study

Exclusion Criteria

1. Inability to give informed consent.
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the subject.
3. Specific exclusions:

   1. Hepatitis B or C
   2. HIV
   3. Abnormal AST or ALT at screening (defined as >/+2x ULN)
4. History of colon cancer in the past two years, or treatment for other cancers within the last 6 months.
5. Investigational drug within one month of treatment
6. Pregnant or breast feeding or trying to become pregnant.
7. Presence of a rectovaginal or perineal body fistula
8. Change in Crohn's immunosuppressive regimen within the 2 months prior to enrollment
9. Uncontrolled intestinal Crohn's disease which will require escalation for medical therapy or surgery within 2 months of enrollment
10. Severe anal canal disease that is stenotic and requires dilation
11. Female participant unwilling to agree to use acceptable contraception methods during participation in study

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events | Month 3
  Number of participants with treatment related adverse events post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease as assessed by protocol
Treatment related adverse events | Month 12
  Number of participants with treatment related adverse events post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease as assessed by protocol

SECONDARY OUTCOMES:
Complete clinical healing | Month 3
  Number of participants with complete clinical healing post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease.
  Complete Healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 3 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical Healing: 100% cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
Complete clinical healing | Month 12
  Number of participants with complete clinical healing post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease.
  Complete Healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 3 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical Healing: 100% cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
Partial clinical healing | Month 3
  Number of participants with partial clinical healing post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease
  Partial clinical healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 2 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical healing: Greater than or equal to 50 % cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
Partial clinical healing | Month 12
  Number of participants with partial clinical healing post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease
  Partial clinical healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 2 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical healing: Greater than or equal to 50 % cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
Lack of response | Month 3
  Number of participants with lack of response post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease
  Lack of response is defined as:
  Radiographic and Clinical healing which does not meet the threshold for Partial Healing
Lack of response | Month 12
  Number of participants with lack of response post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease
  Lack of response is defined as:
  Radiographic and Clinical healing which does not meet the threshold for Partial Healing
Worsening of disease | Month 3
  Number of participants with worsening of disease post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease
  Worsening disease is defined as:
  Radiographic: MRI with a fluid collection >2 cm in 2 of 3 dimensions, edema, inflammation or sign of active inflammatory response. An increased number of tracts may be seen, or increased branching from the primary tract,
  Clinical: Increased drainage per patient report and on clinical exam
Worsening of disease | Month 12
  Number of participants with worsening of disease post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of perianal fistula(s) in the setting of Crohn's disease
  Worsening disease is defined as:
  Radiographic: MRI with a fluid collection >2 cm in 2 of 3 dimensions, edema, inflammation or sign of active inflammatory response. An increased number of tracts may be seen, or increased branching from the primary tract,
  Clinical: Increased drainage per patient report and on clinical exam

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lightner, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Hellers G, Bergstrand O, Ewerth S, Holmstrom B. Occurrence and outcome after primary treatment of anal fistulae in Crohn's disease. Gut. 1980 Jun;21(6):525-7. doi: 10.1136/gut.21.6.525. PMID 7429313
- [Background] Kasparek MS, Glatzle J, Temeltcheva T, Mueller MH, Koenigsrainer A, Kreis ME. Long-term quality of life in patients with Crohn's disease and perianal fistulas: influence of fecal diversion. Dis Colon Rectum. 2007 Dec;50(12):2067-74. doi: 10.1007/s10350-007-9006-5. PMID 17680311
- [Background] Sandborn WJ, Fazio VW, Feagan BG, Hanauer SB; American Gastroenterological Association Clinical Practice Committee. AGA technical review on perianal Crohn's disease. Gastroenterology. 2003 Nov;125(5):1508-30. doi: 10.1016/j.gastro.2003.08.025. No abstract available. PMID 14598268
- [Background] Schwartz DA, Loftus EV Jr, Tremaine WJ, Panaccione R, Harmsen WS, Zinsmeister AR, Sandborn WJ. The natural history of fistulizing Crohn's disease in Olmsted County, Minnesota. Gastroenterology. 2002 Apr;122(4):875-80. doi: 10.1053/gast.2002.32362. PMID 11910338
- [Background] Chaparro M, Zanotti C, Burgueno P, Vera I, Bermejo F, Marin-Jimenez I, Yela C, Lopez P, Martin MD, Taxonera C, Botella B, Pajares R, Ponferrada A, Calvo M, Algaba A, Perez L, Casis B, Mate J, Orofino J, Lara N, Garcia-Losa M, Badia X, Gisbert JP. Health care costs of complex perianal fistula in Crohn's disease. Dig Dis Sci. 2013 Dec;58(12):3400-6. doi: 10.1007/s10620-013-2830-7. Epub 2013 Sep 13. PMID 24026400
- [Background] Aguilera-Castro L, Ferre-Aracil C, Garcia-Garcia-de-Paredes A, Rodriguez-de-Santiago E, Lopez-Sanroman A. Management of complex perianal Crohn's disease. Ann Gastroenterol. 2017;30(1):33-44. doi: 10.20524/aog.2016.0099. Epub 2016 Oct 27. PMID 28042236
- [Background] Adler J, Dong S, Eder SJ, Dombkowski KJ; ImproveCareNow Pediatric IBD Learning Health System. Perianal Crohn Disease in a Large Multicenter Pediatric Collaborative. J Pediatr Gastroenterol Nutr. 2017 May;64(5):e117-e124. doi: 10.1097/MPG.0000000000001447. PMID 27801750
- [Background] Kugathasan S, Judd RH, Hoffmann RG, Heikenen J, Telega G, Khan F, Weisdorf-Schindele S, San Pablo W Jr, Perrault J, Park R, Yaffe M, Brown C, Rivera-Bennett MT, Halabi I, Martinez A, Blank E, Werlin SL, Rudolph CD, Binion DG; Wisconsin Pediatric Inflammatory Bowel Disease Alliance. Epidemiologic and clinical characteristics of children with newly diagnosed inflammatory bowel disease in Wisconsin: a statewide population-based study. J Pediatr. 2003 Oct;143(4):525-31. doi: 10.1067/s0022-3476(03)00444-x. PMID 14571234
- [Background] Markowitz J, Grancher K, Rosa J, Simpser E, Aiges H, Daum F. Highly destructive perianal disease in children with Crohn's disease. J Pediatr Gastroenterol Nutr. 1995 Aug;21(2):149-53. doi: 10.1097/00005176-199508000-00005. PMID 7472900
- [Background] Vernier-Massouille G, Balde M, Salleron J, Turck D, Dupas JL, Mouterde O, Merle V, Salomez JL, Branche J, Marti R, Lerebours E, Cortot A, Gower-Rousseau C, Colombel JF. Natural history of pediatric Crohn's disease: a population-based cohort study. Gastroenterology. 2008 Oct;135(4):1106-13. doi: 10.1053/j.gastro.2008.06.079. Epub 2008 Jul 3. PMID 18692056
- [Background] Kappelman MD, Moore KR, Allen JK, Cook SF. Recent trends in the prevalence of Crohn's disease and ulcerative colitis in a commercially insured US population. Dig Dis Sci. 2013 Feb;58(2):519-25. doi: 10.1007/s10620-012-2371-5. Epub 2012 Aug 29. PMID 22926499